CLINICAL TRIAL: NCT05877196
Title: Precision Medicine in Alzheimer's Disease: A SMART Trial of Adaptive Exercises and Their Mechanisms of Action Using AT(N) Biomarkers to Optimize Aerobic-Fitness Responses (The FIT-AD SMART Trial)
Brief Title: A SMART Trial of Adaptive Exercises to Optimize Aerobic-Fitness Responses
Acronym: SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Banner Alzheimer's Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00017678
Record Dates: First submitted 2023-04-03; First posted 2023-05-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Cognitive Impairment; Cognitive Decline; Memory Loss; Memory Impairment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Memory Disorders | interventions — Exercise; Range of Motion, Articular; Pliability; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Sequential, Multiple Assignment, Randomized Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate Intensity Continuous Training (MICT) (Experimental): Cycling on recumbent stationary cycle at moderate intensity for 30-50 minutes, 3 times per week for 3-6 months
  Interventions: Behavioral: Moderate Intensity Continuous Training (MICT)
- Chair-based Stretch (Sham Comparator): Stretching at low intensity for 30-50 minutes, 3 times per week for 6 months
  Interventions: Behavioral: Chair-based Stretch
- High-Intensity Interval Training (HIIT) (Active Comparator): MICT for 3 months, and then cycling on recumbent stationary cycle at alternate high and moderate intensity for 40 minutes, 3 times per week for 3 months.
  Interventions: Behavioral: High-Intensity Interval Training (HIIT)
- Combined Aerobic Resistance Exercise (CARE) (Active Comparator): MICT for 3 months, and then cycling on recumbent stationary cycle at moderate intensity for 30 minutes, followed by 20-minute strength-building exercise, 3 times per week for 3 months.
  Interventions: Behavioral: Combined Aerobic Resistance Exercise (CARE)

INTERVENTIONS:
Behavioral: Moderate Intensity Continuous Training (MICT) — Aerobic cycling at a moderate intensity (50-75% of heart rate reserve) for 30-50 minutes, 3 times per week for 3-6 months.
  Other Names: Continuous Training; Aerobic exercise; Cardio
  Arms: Moderate Intensity Continuous Training (MICT)
Behavioral: Chair-based Stretch — Stretching while seated for 30-50 minutes, 3 times per week for 6 months.
  Other Names: Stretch; Range of motion; flexibility
  Arms: Chair-based Stretch
Behavioral: High-Intensity Interval Training (HIIT) — Aerobic cycling at a vigorous intensity (80-90% of heart rate reserve 4-minute bouts with 4-minute recovery intervals) for 40 minutes, 3 times per week for 3 months.
  Other Names: HIIT; Vigorous training; Hard exercise
  Arms: High-Intensity Interval Training (HIIT)
Behavioral: Combined Aerobic Resistance Exercise (CARE) — 6 full-body strength-building exercises followed by 30 minutes of MICT cycling (described above). Total duration is 60 minutes, 3 times per week for 3 months.
  Other Names: Strength and Cardio Training; CARE; Combination training; Exercise training
  Arms: Combined Aerobic Resistance Exercise (CARE)

SUMMARY:
The goal of this clinical trial is to test 6 months of aerobic exercise in older adults who are 65 years or older and have mild cognitive impairment (MCI) or probable/possible mild Alzheimer's Disease. The main questions it aims to answer are:

* test the effects of aerobic exercise on aerobic fitness, white matter hyperintensity (WMH) volume, and patient-centered outcomes;
* identify the best exercise to improve aerobic fitness and reduce non-responses over 6 months; and
* examines the mechanisms of aerobic exercise's action on memory in older adults with early AD.

Participants will receive 6 months of supervised exercise, undergo cognitive data collection and exercise testing 5 times over a year span, have an MRI brain scan 3 times over a one-year span, and have monthly follow-up discussions on health and wellness.

DETAILED DESCRIPTION:
The purpose of this Phase II, mechanistic Sequential, Multiple Assignment, Randomized Trial (SMART) is to test the effects of 6-month aerobic exercise on aerobic fitness and MRI and plasma biomarkers in community-dwelling older adults with early Alzheimer's disease (AD). The aims are to (I) test the effects of aerobic exercise on aerobic fitness, white matter hyperintensity (WMH) volume, and patient-centered outcomes; (II) identify the best exercise to improve aerobic fitness and reduce non-responses over 6 months; and (III) examines the mechanisms of aerobic exercise's action on memory in older adults with early AD. This trial builds on our previous work showing inter-individual differences in VO2peak responses to moderate-intensity continuous training (MICT); an ability of plasma neurofilament light chain (NfL) to predict cognition; and 6-month MICT maintained memory, reduced WMH, affected plasma p-tau181, and improved physical function, QoL, and caregiver distress. Aerobic exercise is a promising treatment for Alzheimer's disease (AD) and AD-related dementia (ADRD) but has shown mixed effects on cognition, physical function, behavioral and psychological symptoms of dementia (BPSD), quality of life (QoL), and caregiver burden. These findings are likely due to inter-individual differences in aerobic fitness responses, which have long been established in adults using VO2peak and were first reported in AD/ADRD by our team. Most AD/ADRD exercise trials did not measure VO2peak and those that reported large inter-individual differences in VO2peak responses to MICT. Mechanistically, animal studies support aerobic exercise modifying AD's ATN biomarkers (Amyloid-beta [Aβ], Tau, and Neurodegeneration), but human studies are few and have conflicting findings. Hence, precision exercise is critical to improving VO2peak responses with alternative interventions (high-intensity interval training (HIIT) or combined aerobic & resistance exercise (CARE)). Because VO2peak can improve and peak from 3 months of MICT, 3 months is an ideal time to identify MICT non-responders and initiate HIIT or CARE.

ELIGIBILITY:
Inclusion Criteria:

Participants:

* Clinical diagnosis of MCI or probable and possible mild AD dementia according to 2011 Alzheimer's association-NIA criteria.
* Community-dwelling, e.g., homes and assisted living
* Age 65 years and older
* Medical clearance from PCP or cardiovascular provider
* Have a qualified study partner
* Agree to the blood draws
* Verified MRI safety

Study Partner:

* Age 18 or older
* Contact with participant ≥ 2 times per week for ≥ 6 months
* Know the participant's memory status and ability to perform activities of daily living
* Consent to participant

Exclusion Criteria:

Participants

* Resting HR ≤ 50 or ≥ 100 beats/min after 5-minutes of quiet resting
* American College of Sports Medicine contraindications to exercise
* New, unevaluated symptoms or diseases a healthcare provider has not evaluated
* Abnormal cardiac condition uncovered during VO2peak testing
* Enrollment in another intervention that aims at improving cognition
* Moderate to strenuous exercise ≥150 minutes a week in the previous 6 months
* ≥ 2 anti-depression medications, or poorly managed or unstable depression
* Poorly managed or unstable anxiety

Study partners:

* none

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption | measured at 0 and 6 months
  VO2peak will be assessed from the symptom-limited peak cycle-ergometer test
White Matter Hyperintensity volume | measured at 0 and 6 months
  WMH will be assessed from MRI.

SECONDARY OUTCOMES:
Memory | measured at 0, 6, and 12 months
  Wechsler Memory Scale - Revised; Logical Memory; score 0-50; higher scores indicate less impairment
Physical function | measured at 0, 3, 6, 9, & 12 months
  Short Physical Performance Battery: score 0-12; lower scores indicate poorer physical function
Behavioral and psychiatric symptoms of dementia (BPSD) | measured at 1, 3, 6, 9, & 12 months
  Neuropsychiatric Inventory Questionnaire; symptoms present, if yes, then severity and caregiver distress are reported.
Caregiver burden | measured at 1, 3, 6, 9, & 12 months
  4-item Zarit Burden Interview: score 0-16; higher scores reflect greater burden
Quality of Life (QoL) | measured at 1, 3, 6, 9, & 12 months
  Quality of Life - AD: score 0-52; higher scores reflect greater life satisfaction
Blood amyloid-beta 42 and 40 | measured at 1, 3, 6, 9, & 12 months
  20 mL blood sample collection
Blood phosphorylated tau 181 | measured at 1, 3, 6, 9, & 12 months
  20 mL blood sample collection
Blood total tau, neurofilament light chain | measured at 1, 3, 6, 9, & 12 months
  20 mL blood sample collection

OTHER OUTCOMES:
Dementia severity | measured at 0, 3, 6, 9, & 12 months
  Montreal cognitive Assessment: score 0-30; higher scores reflect less impairment
Executive function | measured at 0, 3, 6, 9, & 12 months
  Trail Making Test: number of seconds required to complete the task; therefore, higher scores reveal greater impairment
Visuospatial ability | measured at 0, 3, 6, 9, & 12 months
  Benson Complex Figure: score 0-17; higher scores reflect better visuospatial abilities.
Language preservation | measured at 0, 3, 6, 9, & 12 months
  Multilingual naming test: count the number of items correctly named; higher counts reflect better language preservation
Fall risk | measured at 0, 3, 6, 9, & 12 months
  Timed up and Go: 3-meter course timed; time recorded in seconds; less time reflects lower fall risk
Social interaction | measured at 0, 3, 6, 9, & 12 months
  Engagement and Independence in Dementia Questionnaire: Scale - not true at all = 0, rarely true = 1, sometimes true = 2, often true = 3, true nearly all of the time = 4; higher ratings reflect more social interaction
Anxiety | measured at 0, 3, 6, 9, & 12 months
  Generalized Anxiety Disorder - 7: 0-21; lower scores reflect less anxiety
Depression | measured at 0, 3, 6, 9, & 12 months
  Geriatric Depression Scale: Score 1-15, lowers scores reflect less depression

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yu, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will create a de-identified dataset and de-identified bio-samples to share at the time of publishing the primary results of our trial or within 9 months of database lock, whichever comes first. The data to be shared include but not limited to:
  * de-identified health history and covariate scores
  * de-identified instrument item and total scores of primary and secondary outcomes
  * de-identified exercise session report data
  * de-identified bio-samples
Time Frame: May 2027
Access Criteria: * a commitment to using the data only for research purposes and not to identify an individual participant
  * a commitment to securing the data using appropriate computer technology
  * a commitment to destroying or returning the data after analyses are completed
  * all data sharing requests must be reviewed and approved by the PI

REFERENCES:
- [Background] Almirall D, Nahum-Shani I, Sherwood NE, Murphy SA. Introduction to SMART designs for the development of adaptive interventions: with application to weight loss research. Transl Behav Med. 2014 Sep;4(3):260-74. doi: 10.1007/s13142-014-0265-0. PMID 25264466
- [Background] Salisbury D, Mathiason MA, Yu F. Exercise Dose and Aerobic Fitness Response in Alzheimer's Dementia: Findings from the FIT-AD Trial. Int J Sports Med. 2022 Sep;43(10):850-858. doi: 10.1055/a-1639-2307. Epub 2021 Sep 7. PMID 34492709
- [Background] Pandey A, Swift DL, McGuire DK, Ayers CR, Neeland IJ, Blair SN, Johannsen N, Earnest CP, Berry JD, Church TS. Metabolic Effects of Exercise Training Among Fitness-Nonresponsive Patients With Type 2 Diabetes: The HART-D Study. Diabetes Care. 2015 Aug;38(8):1494-501. doi: 10.2337/dc14-2378. Epub 2015 Jun 17. PMID 26084342
- [Background] Huang G, Wang R, Chen P, Huang SC, Donnelly JE, Mehlferber JP. Dose-response relationship of cardiorespiratory fitness adaptation to controlled endurance training in sedentary older adults. Eur J Prev Cardiol. 2016 Mar;23(5):518-29. doi: 10.1177/2047487315582322. Epub 2015 Apr 21. PMID 25901000
- [Background] Salisbury D, Yu F. Establishing Reference Cardiorespiratory Fitness Parameters in Alzheimer's Disease. Sports Med Int Open. 2020 Jan 30;4(1):E1-E7. doi: 10.1055/a-1089-4957. eCollection 2020 Jan. PMID 32010759
- [Background] Gomes-Neto M, Duraes AR, Conceicao LSR, Roever L, Silva CM, Alves IGN, Ellingsen O, Carvalho VO. Effect of combined aerobic and resistance training on peak oxygen consumption, muscle strength and health-related quality of life in patients with heart failure with reduced left ventricular ejection fraction: a systematic review and meta-analysis. Int J Cardiol. 2019 Oct 15;293:165-175. doi: 10.1016/j.ijcard.2019.02.050. Epub 2019 Jun 24. PMID 31345646
- [Background] Lee J, Lee R, Stone AJ. Combined Aerobic and Resistance Training for Peak Oxygen Uptake, Muscle Strength, and Hypertrophy After Coronary Artery Disease: a Systematic Review and Meta-Analysis. J Cardiovasc Transl Res. 2020 Aug;13(4):601-611. doi: 10.1007/s12265-019-09922-0. Epub 2019 Oct 27. PMID 31656988
- [Background] Lee J, Stone AJ. Combined Aerobic and Resistance Training for Cardiorespiratory Fitness, Muscle Strength, and Walking Capacity after Stroke: A Systematic Review and Meta-Analysis. J Stroke Cerebrovasc Dis. 2020 Jan;29(1):104498. doi: 10.1016/j.jstrokecerebrovasdis.2019.104498. Epub 2019 Nov 13. PMID 31732460
- [Background] Hautala AJ, Makikallio TH, Kiviniemi A, Laukkanen RT, Nissila S, Huikuri HV, Tulppo MP. Cardiovascular autonomic function correlates with the response to aerobic training in healthy sedentary subjects. Am J Physiol Heart Circ Physiol. 2003 Oct;285(4):H1747-52. doi: 10.1152/ajpheart.00202.2003. Epub 2003 Jun 19. PMID 12816748
- [Background] Burns JM, Johnson DK, Watts A, Swerdlow RH, Brooks WM. Reduced lean mass in early Alzheimer disease and its association with brain atrophy. Arch Neurol. 2010 Apr;67(4):428-33. doi: 10.1001/archneurol.2010.38. PMID 20385908
- [Background] Sugimoto T, Ono R, Murata S, Saji N, Matsui Y, Niida S, Toba K, Sakurai T. Prevalence and associated factors of sarcopenia in elderly subjects with amnestic mild cognitive impairment or Alzheimer disease. Curr Alzheimer Res. 2016;13(6):718-26. doi: 10.2174/1567205013666160211124828. PMID 26863996
- [Background] Karlsen T, Aamot IL, Haykowsky M, Rognmo O. High Intensity Interval Training for Maximizing Health Outcomes. Prog Cardiovasc Dis. 2017 Jun-Jul;60(1):67-77. doi: 10.1016/j.pcad.2017.03.006. Epub 2017 Apr 3. PMID 28385556
- [Background] Levinger I, Shaw CS, Stepto NK, Cassar S, McAinch AJ, Cheetham C, Maiorana AJ. What Doesn't Kill You Makes You Fitter: A Systematic Review of High-Intensity Interval Exercise for Patients with Cardiovascular and Metabolic Diseases. Clin Med Insights Cardiol. 2015 Jun 25;9:53-63. doi: 10.4137/CMC.S26230. eCollection 2015. PMID 26157337
- [Background] Bossers WJ, van der Woude LH, Boersma F, Hortobagyi T, Scherder EJ, van Heuvelen MJ. A 9-Week Aerobic and Strength Training Program Improves Cognitive and Motor Function in Patients with Dementia: A Randomized, Controlled Trial. Am J Geriatr Psychiatry. 2015 Nov;23(11):1106-16. doi: 10.1016/j.jagp.2014.12.191. Epub 2015 Jan 3. PMID 25648055
- [Background] Yu F, Vock DM, Zhang L, Salisbury D, Nelson NW, Chow LS, Smith G, Barclay TR, Dysken M, Wyman JF. Cognitive Effects of Aerobic Exercise in Alzheimer's Disease: A Pilot Randomized Controlled Trial. J Alzheimers Dis. 2021;80(1):233-244. doi: 10.3233/JAD-201100. PMID 33523004
- [Background] Bouchard C, Rankinen T. Individual differences in response to regular physical activity. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S446-51; discussion S452-3. doi: 10.1097/00005768-200106001-00013. PMID 11427769
- [Background] Yu F, Mathiason MA, Han S, Gunter JL, Jones D, Botha H, Jack C Jr. Mechanistic Effects of Aerobic Exercise in Alzheimer's Disease: Imaging Findings From the Pilot FIT-AD Trial. Front Aging Neurosci. 2021 Oct 7;13:703691. doi: 10.3389/fnagi.2021.703691. eCollection 2021. PMID 34690736
- [Background] Yu F, Han SY, Salisbury D, Pruzin JJ, Geda Y, Caselli RJ, Li D. Feasibility and preliminary effects of exercise interventions on plasma biomarkers of Alzheimer's disease in the FIT-AD trial: a randomized pilot study in older adults with Alzheimer's dementia. Pilot Feasibility Stud. 2022 Dec 2;8(1):243. doi: 10.1186/s40814-022-01200-2. PMID 36461134
- [Background] Association As. 2021 Alzheimer's disease facts and figures. Accessed April 21, 2021, 2021. https://www.alz.org/media/Documents/alzheimers-facts-and-figures-infographic.pdf
- [Background] McCleery J, Quinn TJ. Aducanumab and the certainty of evidence. Age Ageing. 2021 Nov 10;50(6):1899-1900. doi: 10.1093/ageing/afab167. No abstract available. PMID 34405228
- [Background] Forbes D, Forbes SC, Blake CM, Thiessen EJ, Forbes S. Exercise programs for people with dementia. Cochrane Database Syst Rev. 2015 Apr 15;2015(4):CD006489. doi: 10.1002/14651858.CD006489.pub4. PMID 25874613
- [Background] Toots A, Littbrand H, Bostrom G, Hornsten C, Holmberg H, Lundin-Olsson L, Lindelof N, Nordstrom P, Gustafson Y, Rosendahl E. Effects of Exercise on Cognitive Function in Older People with Dementia: A Randomized Controlled Trial. J Alzheimers Dis. 2017;60(1):323-332. doi: 10.3233/JAD-170014. PMID 28800328
- [Background] Morris JK, Vidoni ED, Johnson DK, Van Sciver A, Mahnken JD, Honea RA, Wilkins HM, Brooks WM, Billinger SA, Swerdlow RH, Burns JM. Aerobic exercise for Alzheimer's disease: A randomized controlled pilot trial. PLoS One. 2017 Feb 10;12(2):e0170547. doi: 10.1371/journal.pone.0170547. eCollection 2017. PMID 28187125
- [Background] Hoffmann K, Sobol NA, Frederiksen KS, Beyer N, Vogel A, Vestergaard K, Braendgaard H, Gottrup H, Lolk A, Wermuth L, Jacobsen S, Laugesen LP, Gergelyffy RG, Hogh P, Bjerregaard E, Andersen BB, Siersma V, Johannsen P, Cotman CW, Waldemar G, Hasselbalch SG. Moderate-to-High Intensity Physical Exercise in Patients with Alzheimer's Disease: A Randomized Controlled Trial. J Alzheimers Dis. 2016;50(2):443-53. doi: 10.3233/JAD-150817. PMID 26682695
- [Background] van Uffelen JG, Chin A Paw MJ, Hopman-Rock M, van Mechelen W. The effects of exercise on cognition in older adults with and without cognitive decline: a systematic review. Clin J Sport Med. 2008 Nov;18(6):486-500. doi: 10.1097/JSM.0b013e3181845f0b. PMID 19001882
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Smith PJ, Blumenthal JA, Hoffman BM, Cooper H, Strauman TA, Welsh-Bohmer K, Browndyke JN, Sherwood A. Aerobic exercise and neurocognitive performance: a meta-analytic review of randomized controlled trials. Psychosom Med. 2010 Apr;72(3):239-52. doi: 10.1097/PSY.0b013e3181d14633. Epub 2010 Mar 11. PMID 20223924
- [Background] Cancela JM, Ayan C, Varela S, Seijo M. Effects of a long-term aerobic exercise intervention on institutionalized patients with dementia. J Sci Med Sport. 2016 Apr;19(4):293-8. doi: 10.1016/j.jsams.2015.05.007. Epub 2015 Jun 4. PMID 26087884
- [Background] Yang SY, Shan CL, Qing H, Wang W, Zhu Y, Yin MM, Machado S, Yuan TF, Wu T. The Effects of Aerobic Exercise on Cognitive Function of Alzheimer's Disease Patients. CNS Neurol Disord Drug Targets. 2015;14(10):1292-7. doi: 10.2174/1871527315666151111123319. PMID 26556080
- [Background] Arcoverde C, Deslandes A, Moraes H, Almeida C, Araujo NB, Vasques PE, Silveira H, Laks J. Treadmill training as an augmentation treatment for Alzheimer's disease: a pilot randomized controlled study. Arq Neuropsiquiatr. 2014 Mar;72(3):190-6. doi: 10.1590/0004-282X20130231. PMID 24676435
- [Background] Ohman H, Savikko N, Strandberg TE, Kautiainen H, Raivio MM, Laakkonen ML, Tilvis R, Pitkala KH. Effects of Exercise on Cognition: The Finnish Alzheimer Disease Exercise Trial: A Randomized, Controlled Trial. J Am Geriatr Soc. 2016 Apr;64(4):731-8. doi: 10.1111/jgs.14059. Epub 2016 Apr 1. PMID 27037872
- [Background] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Background] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Plymate SR, Fishel MA, Watson GS, Cholerton BA, Duncan GE, Mehta PD, Craft S. Effects of aerobic exercise on mild cognitive impairment: a controlled trial. Arch Neurol. 2010 Jan;67(1):71-9. doi: 10.1001/archneurol.2009.307. PMID 20065132
- [Background] Hernandez SS, Coelho FG, Gobbi S, Stella F. [Effects of physical activity on cognitive functions, balance and risk of falls in elderly patients with Alzheimer's dementia]. Rev Bras Fisioter. 2010 Jan-Feb;14(1):68-74. Portuguese. PMID 20414564
- [Background] Zieschang T, Schwenk M, Becker C, Uhlmann L, Oster P, Hauer K. Falls and Physical Activity in Persons With Mild to Moderate Dementia Participating in an Intensive Motor Training: Randomized Controlled Trial. Alzheimer Dis Assoc Disord. 2017 Oct-Dec;31(4):307-314. doi: 10.1097/WAD.0000000000000201. PMID 28628488
- [Background] Padala KP, Padala PR, Lensing SY, Dennis RA, Bopp MM, Roberson PK, Sullivan DH. Home-Based Exercise Program Improves Balance and Fear of Falling in Community-Dwelling Older Adults with Mild Alzheimer's Disease: A Pilot Study. J Alzheimers Dis. 2017;59(2):565-574. doi: 10.3233/JAD-170120. PMID 28655135
- [Background] Toots A, Littbrand H, Lindelof N, Wiklund R, Holmberg H, Nordstrom P, Lundin-Olsson L, Gustafson Y, Rosendahl E. Effects of a High-Intensity Functional Exercise Program on Dependence in Activities of Daily Living and Balance in Older Adults with Dementia. J Am Geriatr Soc. 2016 Jan;64(1):55-64. doi: 10.1111/jgs.13880. PMID 26782852
- [Background] Bossers WJ, van der Woude LH, Boersma F, Hortobagyi T, Scherder EJ, van Heuvelen MJ. Comparison of Effect of Two Exercise Programs on Activities of Daily Living in Individuals with Dementia: A 9-Week Randomized, Controlled Trial. J Am Geriatr Soc. 2016 Jun;64(6):1258-66. doi: 10.1111/jgs.14160. PMID 27321604
- [Background] Telenius EW, Engedal K, Bergland A. Effect of a high-intensity exercise program on physical function and mental health in nursing home residents with dementia: an assessor blinded randomized controlled trial. PLoS One. 2015 May 14;10(5):e0126102. doi: 10.1371/journal.pone.0126102. eCollection 2015. PMID 25974049
- [Background] Suttanon P, Hill KD, Said CM, Williams SB, Byrne KN, LoGiudice D, Lautenschlager NT, Dodd KJ. Feasibility, safety and preliminary evidence of the effectiveness of a home-based exercise programme for older people with Alzheimer's disease: a pilot randomized controlled trial. Clin Rehabil. 2013 May;27(5):427-38. doi: 10.1177/0269215512460877. Epub 2012 Nov 1. PMID 23117349
- [Background] Sobol NA, Hoffmann K, Frederiksen KS, Vogel A, Vestergaard K, Braendgaard H, Gottrup H, Lolk A, Wermuth L, Jakobsen S, Laugesen L, Gergelyffy R, Hogh P, Bjerregaard E, Siersma V, Andersen BB, Johannsen P, Waldemar G, Hasselbalch SG, Beyer N. Effect of aerobic exercise on physical performance in patients with Alzheimer's disease. Alzheimers Dement. 2016 Dec;12(12):1207-1215. doi: 10.1016/j.jalz.2016.05.004. Epub 2016 Jun 23. PMID 27344641
- [Background] Lam FM, Huang MZ, Liao LR, Chung RC, Kwok TC, Pang MY. Physical exercise improves strength, balance, mobility, and endurance in people with cognitive impairment and dementia: a systematic review. J Physiother. 2018 Jan;64(1):4-15. doi: 10.1016/j.jphys.2017.12.001. Epub 2017 Dec 27. PMID 29289581
- [Background] Rodrigues SLDS, Silva JMD, Oliveira MCC, Santana CMF, Carvalho KM, Barbosa BJAP. Physical exercise as a non-pharmacological strategy for reducing behavioral and psychological symptoms in elderly with mild cognitive impairment and dementia: a systematic review of randomized clinical trials. Arq Neuropsiquiatr. 2021 Dec;79(12):1129-1137. doi: 10.1590/0004-282X-ANP-2020-0539. PMID 34877985
- [Background] Fleiner T, Leucht S, Forstl H, Zijlstra W, Haussermann P. Effects of Short-Term Exercise Interventions on Behavioral and Psychological Symptoms in Patients with Dementia: A Systematic Review. J Alzheimers Dis. 2017;55(4):1583-1594. doi: 10.3233/JAD-160683. PMID 27911304
- [Background] Heesterbeek M, Van der Zee EA, van Heuvelen MJG. Passive exercise to improve quality of life, activities of daily living, care burden and cognitive functioning in institutionalized older adults with dementia - a randomized controlled trial study protocol. BMC Geriatr. 2018 Aug 14;18(1):182. doi: 10.1186/s12877-018-0874-4. PMID 30107789
- [Background] Song D, Yu DSF. Effects of a moderate-intensity aerobic exercise programme on the cognitive function and quality of life of community-dwelling elderly people with mild cognitive impairment: A randomised controlled trial. Int J Nurs Stud. 2019 May;93:97-105. doi: 10.1016/j.ijnurstu.2019.02.019. Epub 2019 Mar 5. PMID 30901716
- [Background] Holthoff VA, Marschner K, Scharf M, Steding J, Meyer S, Koch R, Donix M. Effects of physical activity training in patients with Alzheimer's dementia: results of a pilot RCT study. PLoS One. 2015 Apr 17;10(4):e0121478. doi: 10.1371/journal.pone.0121478. eCollection 2015. PMID 25884637
- [Background] Yu F, Nelson NW, Savik K, Wyman JF, Dysken M, Bronas UG. Affecting cognition and quality of life via aerobic exercise in Alzheimer's disease. West J Nurs Res. 2013 Jan;35(1):24-38. doi: 10.1177/0193945911420174. Epub 2011 Sep 12. PMID 21911546
- [Background] Lortie G, Simoneau JA, Hamel P, Boulay MR, Landry F, Bouchard C. Responses of maximal aerobic power and capacity to aerobic training. Int J Sports Med. 1984 Oct;5(5):232-6. doi: 10.1055/s-2008-1025911. PMID 6500788
- [Background] Hecksteden A, Pitsch W, Rosenberger F, Meyer T. Repeated testing for the assessment of individual response to exercise training. J Appl Physiol (1985). 2018 Jun 1;124(6):1567-1579. doi: 10.1152/japplphysiol.00896.2017. Epub 2018 Jan 11. PMID 29357481
- [Background] Karavirta L, Hakkinen K, Kauhanen A, Arija-Blazquez A, Sillanpaa E, Rinkinen N, Hakkinen A. Individual responses to combined endurance and strength training in older adults. Med Sci Sports Exerc. 2011 Mar;43(3):484-90. doi: 10.1249/MSS.0b013e3181f1bf0d. PMID 20689460
- [Background] Robinson MM, Dasari S, Konopka AR, Johnson ML, Manjunatha S, Esponda RR, Carter RE, Lanza IR, Nair KS. Enhanced Protein Translation Underlies Improved Metabolic and Physical Adaptations to Different Exercise Training Modes in Young and Old Humans. Cell Metab. 2017 Mar 7;25(3):581-592. doi: 10.1016/j.cmet.2017.02.009. PMID 28273480
- [Derived] Yu F, Todd M, Salisbury D, Maxfield M, Pruzin J, Joseph RP, Su Y, Li D, Baena E, Coon D. Precision exercise in older adults with early Alzheimer's disease: The study protocol of the FIT-AD Sequential, Multiple Assignment, Randomized Trial (SMART). Trials. 2025 Oct 15;26(1):416. doi: 10.1186/s13063-025-09040-0. PMID 41094623